CLINICAL TRIAL: NCT03890016
Title: Comparing Modified Lee White Method Against 20 Minute Whole Blood Clotting Test as a Bedside Coagulation Test in Snake Envenomation Victims
Brief Title: Study Comparing Modified Lee White Clotting Time Against Twenty Minute Whole Blood Clotting Test in Snakebite Victims
Acronym: LAT
Status: Completed | Type: Observational
Sponsor: Appu Suseel (Other)
Responsible Party: Sponsor-Investigator, Appu Suseel, Assistant Professor, Jubilee Mission Medical College and Research Institute
Organization: Jubilee Mission Medical College and Research Institute (Other)
Other Study IDs: 01/19/IEC/JMMC&RI; U1111-1228-5286 (Other: World Health Organisation)
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Coagulation Defect; Snake Bites
Keywords: Modified Lee and White Method; 20'WBCT; Whole Blood Clotting Test
MeSH Terms: conditions — Hemostatic Disorders; Snake Bites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- snakebite victims: Victims of snakebite presenting to the Emergency Department of Jubilee Mission Medical College and Research Institute
  Interventions: Diagnostic Test: 20'Whole Blood ClottingTest (WBCT); Diagnostic Test: Modified Lee and White (MLW) Method Clotting Time

INTERVENTIONS:
Diagnostic Test: 20'Whole Blood ClottingTest (WBCT) — 1ml of blood drawn from snake bite victims in clean glass test tubes of 1 cm diameter Kept undisturbed for a period of 20 minutes (measured by a stop watch). At the end of 20 minutes the tube is tilted to see if the blood has clotted or not.
  If a well formed clot is not formed, the test is recorded as 'abnormal'.
  If the clot seems well formed, it is further observed for a period of 30 minutes to look for dissolution of the formed clot and would be termed "clot lysis". Clot lysis indicates an unstable clot.
  Other Names: 20'WBCT
Diagnostic Test: Modified Lee and White (MLW) Method Clotting Time — The blood collected in three additional test tubes would be utilised for MLW.
  The three test tubes would be kept on a rack at ambient temperature.
  The blood sample would be drawn in a 5cc syringe and 1 ml would be added in the three test tubes consecutively.
  The test tube would be left undisturbed for 5 minutes, after that the first tube would be tilted approximately to check for clot formation every 30 seconds while the other tubes are left undisturbed.
  After the blood in the first tube has clotted, the time would be noted and the second tube would be tilted every 30 seconds and examined.
  Following its clotting, the third tube would be examined. The time at which the third tube is recorded as the CT value.
  Once clotted, then the sample in the all three test tube would be assessed at 20 minute and 30 min to look for breakup or lysis of the clot.

SUMMARY:
20 minute Whole Blood Clotting Test(20'WBCT) recommended by World Health Organisation guidelines is probably the most routinely employed bed side screening tool in the country.

The Modified Lee and White (MLW) method gives a value which when performed serially gives a trend in clotting time which the investigators hypothesise to be a better tool in serially assessing the victim compared to the 20'WBCT.

The investigators propose that delayed reading of both MLW and 20'WBCT to check for clot stability at 30 minutes also provides added information in management of snake bite victims.

DETAILED DESCRIPTION:
Envenomation by snakes is common in India. Hematotoxic bites cause the highest morbidity and mortality in Kerala, a state in the south of India.

20 minute Whole Blood Clotting Test(20'WBCT) recommended by World Health Organisation guidelines is probably the most routinely employed bed side screening tool in the country. It is the tool of choice due to its cost effectiveness in low and middle income countries (LMIC).

The reliability of 20'WBCT is questionable with respect to not just its rapidity but also its reliability. There is no standardisation for the test and procedure.

Modified Lee White (MLW) Method for coagulation is a cheap bed side test used as part of the standard treatment protocol of snake bite victims. The MLW method gives a value which when performed serially gives a trend in clotting time which the investigators hypothesise to be a better tool in serially assessing the victim compared to the World Health Organisation recommended 20'WBCT.

The investigators also propose that delayed reading of both MLW and 20'WBCT to check for clot stability also provides added information in management of snake bite victims.

The bed side coagulation test done, forms the trigger to commence antivenom in snake bite victims with hematotoxicity in resource limited settings.

Lee White (MLW) Method for coagulation is a test that has been employed for decades to assess coagulation in Jubilee Mission Hospital, Medical College and Research Institute in Thrissur for snake bite victims. It is a cheap bed side test used as part of the standard treatment protocol of snake bite victims. The MLW method gives a value which when performed serially gives a trend in clotting time which the investigators hypothesise to be a better tool in serially assessing the victim compared to the World Health Organisation recommended 20'WBCT.

The investigators also propose that delayed reading of both MLW and 20'WBCT to check for clot stability or 'clot lysis' also provides added information in management of snake bite victims.

ELIGIBILITY:
Inclusion Criteria:

1. All victims of snake bite presenting to the emergency department AND
2. Consenting to be part of the study

Exclusion Criteria:

1. Those not providing a written informed consent OR
2. Those on anticoagulants or antiplatelets OR
3. With a known hematological disorder OR
4. A known history of chronic liver disease OR
5. Received antivenom or blood products following snakebite at another centre

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All snake bite victims presenting to the emergency department of Jubilee mission medical college and research institute.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of serial Modified Lee White Method(MLW) in comparison with twenty minute Whole Blood Clotting Test in detecting coagulopathy in snakebite victims. | 48 hours of snakebite
Sensitivity and Specificity of admission Modified Lee White Method(MLW) and twenty minute Whole Blood Clotting Test in detecting coagulopathy in snakebite victims. | 48 hours
  Comparing MLW and 20'WBCT to gold standard tests like Prothrombin Time (PT) and activated partial thromboplastin time (aPTT)

SECONDARY OUTCOMES:
Sensitivity of admission 20'WBCT and MLW to diagnose Russells viper (Daboia ruselli) envenomation | 48hours
Sensitivity of admission 20'WBCT and MLW to diagnose Hump-nosed pit viper (Hypnale hypnale) envenomation | 48hours
Time to detection of hematotoxic envenomation in MLW and 20'WBCT | 48 hours
Sensitivity and specificity of delayed reading of clotting time and clotting test at 30 minutes in detecting coagulopathy | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Siju Varghese Abraham, M.D, Study Director — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India